CLINICAL TRIAL: NCT05865782
Title: Skolgårdsprojketet: Bygga om skolgårdar i Stockholm Med grönska för Att öka Skolbarns Fysisk Aktivitet Och hälsa Samt Mildra klimatförändringarna i städer
Brief Title: Reconstructing Schoolyards With Greenery to Increase Schoolchildren's Physical Activity and Mitigate Climate Changes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The City of Stockholm (Unknown); Cancerfonden (Unknown); Arwidssonstiftelsen (Unknown)
Responsible Party: Principal Investigator, Daniel Berglind, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: The Schoolyard project
Record Dates: First submitted 2023-03-29; First posted 2023-05-19 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Physical Inactivity; Environmental Exposure; Mental Health Wellness 1
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Study design The current study will be designed as a quasi-experimental stepped-wedge intervention where schools undertaking schoolyard reconstruction will act as both control and intervention schools. Five schools will yearly receive the intervention (schoolyard reconstruction) at 4 different time points (during the summer breaks in 2023, 2024, 2025 and 2026) and the schools not receiving the intervention the specific year will act as control schools. The units where the proposed outcomes will be observed will be 2nd and 5th grade children (individual level) in the participating schools. Each year, a cross-sectional sample of 2nd and 5th grade children will be measured in all participating schools.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Schoolyard reconstruction (Experimental): Schools undertaking schoolyard reconstruction will act as both control and intervention schools. Each year, a cross-sectional sample of 2nd and 5th grade children will be measured in all participating schools.
  Interventions: Behavioral: Schoolyard reconstruction

INTERVENTIONS:
Behavioral: Schoolyard reconstruction — The current study will be designed as a quasi-experimental stepped-wedge intervention where schools undertaking schoolyard reconstruction will act as both control and intervention schools. By using the stepped-wedge study design, with internal control schools, will enable the control for the seasonal variation in children's physical activity levels and for the age-related decline in physical activity throughout childhood. That is, without control schools we would be unable to attribute a change in physical activity to the reconstruction of the schoolyards - as any difference in physical activity before and after the schoolyard reconstruction in the intervention group could be explained by the natural change in physical activity over time.

SUMMARY:
By reconstructing schoolyards with greenery, physical activity levels among children can be increased at the population level and also mitigate health and environmental risks resulting from rising climate changes in urban areas.

The overarching purpose of the proposed project is to:

i. increase physical activity levels among school-aged children, independent of socioeconomic factors, and thus affect short- and long-term health outcomes on a population level ii. establish an evidence-based bottom-up approach for schoolyard reconstructions iii. evaluate the cost-effectiveness of schoolyard reconstructions with greening on health outcomes and its environmental impact

DETAILED DESCRIPTION:
Background More than half of Swedish schoolchildren do not meet the physical activity guidelines, which will have long-lasting effects on their health in adulthood. The school environment plays a crucial role in establishing healthy physical activity behaviors for a population.

A formal decision has been made to reconstruct 15 Stockholm public schoolyards from 2024 to 2026. This project is evaluating the effects of this decision.

Project design The project is designed as a quasi-experimental stepped-wedge trial, with schools serving as both intervention and control schools. Over the course of 3 years (2023-2026), a total of 15 schoolyard reconstructions will be evaluated, with 5 reconstructions per year. The units of observation will be second and fifth grade children, totaling 2,700 children.

Methods for data collection The following primary and secondary outcomes will be measured at baseline (May) and at follow-up one year later (May the following year), in all schools, among participating children.

Research questions

1. How does schoolyard reconstruction affect physical activity levels, blood pressure, BMI, mental health, sleep, and sick leave in schoolchildren?
2. Which components of schoolyard reconstruction are associated with changes (if any) in physical activity levels, blood pressure, BMI, mental health, sleep, and sick leave in schoolchildren?
3. What would be the cost-effectiveness of schoolyard reconstruction on the health outcomes, physical activity levels, blood pressure, BMI, mental health, sleep, and sick leave of school children, as well as its impact on the microclimate and CO2-emissions in urban areas, if the project would be extended to other schools in Stockholm, and possibly Sweden as a whole?

Intervention description and theory The schoolyard reconstruction process will use a participatory bottom-up co-creation development approach involving students, school personnel and researchers and will be evidence-based, using prior knowledge on schoolyard features that are associated with children's physical activity during school-hours. Additionally, the schoolyard reconstruction intervention process will be discussed and acknowledged among all co-creators to increase the engagement, buy-in, feasibility, relevance and sustainability of the schoolyard reconstruction intervention.

Workshops will be held by experts from the City of Stockholm, Karolinska institutet and landscape architects with greenery experience, students, school personnel (e.g., principal, teachers etc.), at each school before schoolyard reconstruction initiation. The workshops will process the design and dimension of what components the schoolyard reconstruction should encompass, reflecting school personnel/students' proposals and local challenges and needs.

Statistical analyses Each school undertaking schoolyard renewal will be treated as an independent unit and analyzed separately (i.e., analyses of five separate schoolyard renewals, with appurtenant intervention school, per year). We will match each intervention school, based on school size and socioeconomic factors, with a control school undertaking schoolyard renewal at a different time-point. We deem it appropriate to analyze each control-intervention pair separately as each intervention school represent a unique schoolyard renewal intervention package (different reconstructions). We will also pool the pair-specific estimates, as appropriate, to quantify a global estimate of the total effect of the project.

Societal relevance Most schoolyards in Stockholm lack appealing play areas and are instead dominated by concrete and asphalt surfaces. As school participation is not segregated by socioeconomic factors, schoolyard reconstructions that promote physical activity can benefit children from all socioeconomic groups. Additionally, reconstructing schoolyards with greenery can mitigate health and environmental risks associated with increasing climate changes in urban areas.

ELIGIBILITY:
Inclusion Criteria:

On school level:

-School selected for schoolyard reconstruction by the City of Stockholm

On individual level (schoolchildren):

* Enrolled in participating school
* 8-13 years old at the time of study start
* In 2nd or 5th grade
* Parents signed informed consent

Exclusion Criteria:

On school level:

-School not selected for schoolyard reconstruction by the City of Stockholm

On individual level (schoolchildren):

* Not enrolled in participating school
* Outside 8-13 years old age range and/or not in 2nd or 5th grade
* Parents declined informed consent

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3600 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity levels in children | 12 months change from baseline (in May before schoolyard reconstruction) to 1-year follow-up (in May 1 year later) in physical activity levels
  Physical activity levels in terms of daily minutes in moderate to vigorous physical activity, total physical activity and daily steps measured objectively by Actigraph GT3X+ accelerometers

SECONDARY OUTCOMES:
Change in musculoskeletal fitness in children | 12 months change from baseline (in May before schoolyard reconstruction) to 1-year follow-up (in May 1 year later) in musculoskeletal fitness (handgrip strength)
  Musculoskeletal fitness, in terms of handgrip strength ,will be measured by an analogue dynamometer (TKK 5825, Grip-A, Takei, Tokyo, Japan).
Change in weight in children | 12 months change from baseline (in May before schoolyard reconstruction) to 1-year follow-up (in May 1 year later) in weight
  Weight (in kilograms) will be measured with validated scales
Change in height in children | 12 months change from baseline (in May before schoolyard reconstruction) to 1-year follow-up (in May 1 year later) in height
  Height (in centimeters) will be measured with validated stadiometers
Change in blood pressure in children | 12 months change from baseline (in May before schoolyard reconstruction) to 1-year follow-up (in May 1 year later) in blood pressure
  Systolic and diastolic blood pressure will be measured three times (and we will use the mean value of the two last measures), in the seated position after a five-minutes rest, using a medically approved automatic digital blood pressure monitor
Change in mental health in children | 12 months change from baseline (in May before schoolyard reconstruction) to 1-year follow-up (in May 1 year later) in mental health
  Psychosocial functioning of children will be assessed by a parental proxy report of the Strength and Difficulty Questionnaire. Total difficulties score is generated by summing scores from all the scales except the prosocial scale and ranges from 0 to 40, higher score means worse outcome
Change in sleep in children | 12 months change from baseline (in May before schoolyard reconstruction) to 1-year follow-up (in May 1 year later) in sleep
  Sleep will be measured objectively by the GT3X+ accelerometer. In addition, parents will answer questions about children's sleep duration and quality in the last 6 months in the sleep questionnaire. These sleep questions are adapted from the validated Ages and Stages Questionnaire. The sleep quality score ranges from 0-12 and higher score means better outcome
Change in sick leave | 12 months change from baseline (in May before schoolyard reconstruction) to 1-year follow-up (in May 1 year later) in sick leave
  Sick leave frequency and duration (occasions and days) will be collected from a Stockholm City database
Change in children's perception of the schoolyard quality | 12 months change from baseline (in May before schoolyard reconstruction) to 1-year follow-up (in May 1 year later) in children's perception of the schoolyard quality
  A questionnaire with 7 items, previously used to evaluate schoolyard reconstructions, will be used to assess children's perception of the schoolyard quality
Schoolyard reconstruction costs | Collected through study completion, an average of 1 year
  Detailed budget costs for each schoolyard reconstruction, e.g., play equipment, construction and maintenance costs will be collected for each separate schoolyard reconstruction and further used for health economic evaluations
Environmental impact of schoolyard reconstruction | Collected through study completion, an average of 1 year
  Based on greenery increase from the schoolyard reconstruction we will use models for impact on CO2-emissions and albedo (Δα) scores (i.e., reflective properties from greenery) as environmental benefit outcomes
Incidents in the schoolyard | Change in number of incidents from 12 months before to 12 months after schoolyard reconstruction
  Number of incidents (e.g., conflicts, sun burns etc.) from before to after schoolyard reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Berglind, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Swedish law do not allow individual data sharing without ethical permission.